CLINICAL TRIAL: NCT02768558
Title: Randomized, Double Blinded Phase III Trial of Cisplatin and Etoposide Plus Thoracic Radiation Therapy Followed By Nivolumab/Placebo For Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Cisplatin and Etoposide Plus Radiation Followed By Nivolumab/Placebo For Locally Advanced NSCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Another treatment found efficacious
Sponsor: RTOG Foundation, Inc. (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RTOG 3505; RF 3505 (Other: RTOG Foundation); CA209-333 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2020-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Cancer; NSCLC; Nivolumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Cisplatin; Etoposide; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nivolumab (Experimental): 60 Gy of radiation therapy given concurrently with cisplatin-etoposide chemotherapy followed by nivolumab
  Interventions: Radiation: Radiation Therapy (RT); Drug: Cisplatin; Drug: Etoposide; Drug: Nivolumab
- Placebo (Placebo Comparator): 60 Gy of radiation therapy given concurrently with cisplatin-etoposide chemotherapy followed by placebo
  Interventions: Radiation: Radiation Therapy (RT); Drug: Cisplatin; Drug: Etoposide; Other: Placebo

INTERVENTIONS:
Radiation: Radiation Therapy (RT) — 2 Gy fractions once a day, 5 days per week, for a total of 60 Gy in 30 fractions.
  Other Names: 3 Dimensional Conformal Radiation Therapy (3DCRT); Intensity Modulated Radiation Therapy (IMRT)
Drug: Cisplatin — Concurrently with radiation therapy, 50 mg/m2, IV, on days 1, 8, 29, and 36, to begin with day 1 of radiation therapy.
  Other Names: Platinol
Drug: Etoposide — Concurrently with radiation, 40 mg/m2, IV, on days 1-5 and 29-33, to begin with day 1 of radiation therapy.
  Other Names: VP-16
Drug: Nivolumab — Beginning 4-12 weeks after chemoradiation, 240 mg, IV, every 2 weeks for 16 weeks, then 480 mg, IV, for 36 weeks.
  Other Names: Opdivo
  Arms: Nivolumab
Other: Placebo — Beginning 4-12 weeks after chemoradiation, 240 mg, IV, every 2 weeks for 16 weeks, then 480 mg, IV, for 36 weeks.
  Arms: Placebo

SUMMARY:
Patients with Stage III unresectable non-small cell lung cancer will receive thoracic radiation, cisplatin and etoposide followed by nivolumab or placebo given every 2 weeks for a year.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the Overall Survival (OS) for patients with Stage III unresectable non-small cell lung cancer treated with or without nivolumab following concurrent chemoradiation.

II. To compare Progression-Free Survival (PFS) according to RECIST 1.1 criteria for patients with Stage III unresectable non-small cell lung cancer treated with or without nivolumab following concurrent chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of non-small cell lung cancer (NSCLC) with unresectable, medically inoperable disease, or patients who refuse resection stage IIIA or stage IIIB disease (AJCC 7th edition)
* History/physical examination within 30 days prior to registration
* Computed tomography (CT) scan with IV contrast (CT scan without contrast acceptable if IV contrast is medically contraindicated) of the lung and upper abdomen through the adrenal glands within 60 days prior to registration (recommended within 30 days prior to registration)
* Magnetic resonance imaging (MRI) of the brain with contrast (or CT with contrast if MRI is medically contraindicated) within 60 days prior to registration; note: the use of intravenous contrast is required for the MRI or CT (unless medically contra-indicated).
* Whole-body fluorodeoxyglucose (FDG)-positron emission tomography (PET)/CT within 60 days prior to registration; Note: patients do not need to have a separate CT of chest and upper abdomen with contrast if PET/CT imaging includes a high quality CT chest with contrast.
* Age ≥ 18 years
* The trial is open to both genders
* Zubrod Performance status of 0-1
* Forced Expiratory Volume at one second (FEV1) > 1.2 liters; Diffusion Capacity of Lung for Carbon Monoxide (DLCO) ≥ 50% predicted
* Patients must be at least 3 weeks from prior thoracotomy (if performed); if prior thoracotomy then measurable disease on imaging must be present
* Negative serum pregnancy test within three days prior to registration for women of childbearing potential
* An archived tumor block or punches instead block must be available for submission for programmed death-ligand 1 (PD-L1) analysis. If an archived tumor block sample cannot be shipped for this study, then two 3mm punches from the core needle biopsy blocks may be provided for analysis. Note: core or excisional biopsy is required for this study. Fine needle aspirates (FNA) and cytology specimens are not adequate for PD-L1 analysis.
* Agreement of women of childbearing potential to use highly effective contraception during receipt of study drug and up to 161 days (23 weeks) from the last dose of nivolumab/placebo and men receiving nivolumab/placebo who are sexually active with women of childbearing potential to use highly effective contraception during receipt of study drug for 31 weeks from the last dose of nivolumab/placebo.

Exclusion Criteria:

* Definitive clinical or radiological evidence of metastatic disease
* Prior or current invasive malignancy (except non-melanomatous skin cancer, localized bladder and prostate cancer) unless disease free for a minimum of 2 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields. For example, patients with prior breast radiotherapy treatments would likely be excluded.
* Prior systemic treatment with and anti-programmed cell death protein 1 (PD1), anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) (antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
* Known immunosuppressive disease, for example HIV infection or history of bone marrow transplant or chronic lymphocytic leukemia (CLL)
* Chronic Obstructive Pulmonary Disease (COPD) exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration. COPD requiring chronic oral steroid therapy
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
* Transmural myocardial infarction within the last 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* History of symptomatic or p previously established interstitial lung disease
* Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection;
* History of severe hypersensitivity reaction to any monoclonal antibody or allergy to study drug components
* As there is potential for hepatic toxicity with nivolumab, drugs with a predisposition to hepatotoxicity should be used with caution in patients treated with nivolumab-containing regimen
* Pregnancy, nursing females or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gerber, MD, Principal Investigator — RTOG Foundation
Locations (16):
- United States (16):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - Mount Sinai Cancer Research Center, Miami Beach, Florida
  - Nancy N. & J.C. Lewis Cancer & Research Pavilion at St. Joseph's/Candler Hospital, Savannah, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Mercy Medical Cancer Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Metro Health Medical Center, Cleveland, Ohio
  - Reading Hospital/McGlinn Cancer Institute, West Reading, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Mason, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerber DE, Urbanic JJ, Langer C, Hu C, Chang IF, Lu B, Movsas B, Jeraj R, Curran WJ, Bradley JD. Treatment Design and Rationale for a Randomized Trial of Cisplatin and Etoposide Plus Thoracic Radiotherapy Followed by Nivolumab or Placebo for Locally Advanced Non-Small-Cell Lung Cancer (RTOG 3505). Clin Lung Cancer. 2017 May;18(3):333-339. doi: 10.1016/j.cllc.2016.10.009. Epub 2016 Oct 26. PMID 27923550

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Registered patients who submitted tissue for PD-L1 assessment and had no evidence of distant metastases or local disease progression at the second step registration were randomized. Of 20 registered patients, 8 were randomized.
Period: Overall Study
Arm/Group | Nivolumab | Placebo
Started | 3 | 5
Eligible (Participants contributing data to results are considered to have completed the study) | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Placebo | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Median (Full Range); unit: years] | 72 [71 to 73] | 64 [57 to 69] | 67.5 [57 to 73]
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 0 | 1 | 1
  60-69 years | 0 | 4 | 4
  ≥ 70 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 0 | 1 | 1
    1 | 3 | 4 | 7
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 2 | 3 | 5
  Squamous cell carcinoma | 1 | 2 | 3
PD-L1 [Count of Participants; unit: Participants] — The programmed death-ligand 1 (PDL1) rate is obtained via analysis of a tissue biopsy and indicates the % of stained cells PD-L1, which is a protein which helps to keep immune cells from targeting healthy cells. Cancer cells may have high quantities of PD-L1 in order to avoid being targeted by the immune system.
  Participants
    < 1% | 0 | 3 | 3
    ≥ 1% | 2 | 1 | 3
    Not Evaluable | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Survival time is defined as time from registration to date of death from any cause and was to be estimated by the Kaplan-Meier method. Given the limited follow-up due to early closure and termination of data collection, only the number of patients last reported to be alive at time of study termination is reported and no statistical testing was done.
Time Frame: From registration to study termination. Maximum follow-up was 14.9 months.
Population: Eligible participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 3 | 5
Participants | 2 | 5

2. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression is defined using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST) guideline v1.1 as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions at any location. Progression was to be determined by an independent radiology review committee using scans submitted to a central location.
  Progression-free survival time is defined as time from registration to the date of first progression, death, or last known follow-up (censored) and was to be estimated by the Kaplan-Meier method.
Time Frame: From registration to study termination. Maximum follow-up was 14.9 months.
Population: Central review of imaging to determine progression was not performed due to early study closure therefore progression (and hence progression-free survival) could not be determined.
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Grade 3+ Adverse Events
Description: Adverse events (AE) are graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From registration to study termination. Maximum follow-up was 14.9 months.
Population: Eligible participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 3 | 5
Participants | 3 | 3

4. Secondary Outcome: Percentage of Participants With Deterioration in Functional Assessment of Cancer Therapy - Trial Outcome Index for Lung Cancer (FACT-TOI) at 15 Months
Description: FACT-TOI is a measure of 21 items that sum the functional well being (FWB), physical well being (PWB), and the lung cancer subscale (LCS) of the Functional Assessment of Cancer Therapy - Lung (FACT-L) QOL instrument, used for measuring QOL in patients with lung cancer. All items are rated on a 5 item (point) Likert Scale, from 0 (not at all) to 4 (very much). FACT-TOI is scored by summing the individual scale scores, with higher scores indicating better quality of life. Deterioration was defined as a decrease of 5 points or more from baseline.
Time Frame: Baseline and 15 months
Population: No participants had a 15-month FACT-TOI assessment
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival by PD-L1 Status
Time Frame: From registration to study termination. Maximum follow-up was 14.9 months.
Population: Data is not reported because the primary endpoints were not determined to have positive results. [Per the protocol, this subgroup analysis was to occur only if either of the primary endpoints were determined to have positive results.]
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progression-Free Survival by PD-L1 Status
Time Frame: From registration to study termination. Maximum follow-up was 14.9 months.
Population: as for outcome 5
Arm/Group | Nivolumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were to be reported every 3 months until 2 years post-chemoradiation, then every 6 months until 5 years post-chemoradiation, then yearly until study termination.
Arm/Group | Nivolumab | Placebo
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=3) | Placebo (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Death NOS (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=3) | Placebo (N=5)
Anemia (Blood and lymphatic system disorders) | 3 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Blurred vision (Eye disorders) | 0 | 1
Eye disorders - Other (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 4
Esophagitis (Gastrointestinal disorders) | 2 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 5
General disorders and administration site conditions - Other (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Immune system disorders - Other (Immune system disorders) | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
Investigations - Other (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 2
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 3 | 1
Serum amylase increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 2 | 1
White blood cell decreased (Investigations) | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Nervous system disorders - Other (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Confusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early due to the reporting of another study which changed this population's standard of care and rendered the control arm obsolete. Eight of the planned 550 analyzable participants were enrolled at the time of termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT02768558/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT02768558/ICF_001.pdf